CLINICAL TRIAL: NCT01067651
Title: Comparison of Two Different Cast Materials for the Treatment of Congenital Idiopathic Clubfoot Using the Ponseti Method: A Prospective Randomized Controlled Trial
Brief Title: Comparison of Casting Materials for the Treatment of Clubfoot Using the Ponseti Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Children's Hospital (Other)
Responsible Party: Dr. Jason Howard, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-20062
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2007-04

CONDITIONS: Clubfoot; Ponseti Method; Talipes Equinovarus; Casting
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plaster of Paris (POP) (Active Comparator)
  Interventions: Device: Plaster of Paris (POP) casting using the Ponseti Method
- semi-rigid fiberglass softcast (SRF, 3M Scotchcast) (Active Comparator)
  Interventions: Device: Semi-Rigid Fiberglass softcast using the Ponseti Method

INTERVENTIONS:
Device: Plaster of Paris (POP) casting using the Ponseti Method
  Arms: Plaster of Paris (POP)
Device: Semi-Rigid Fiberglass softcast using the Ponseti Method
  Arms: semi-rigid fiberglass softcast (SRF, 3M Scotchcast)

SUMMARY:
The purpose of this study was to determine the influence of cast material on correction of congenital idiopathic clubfeet using the Ponseti method.

DETAILED DESCRIPTION:
Congenital idiopathic clubfoot is the most common congenital deformity in children. It can be a major cause of disability for children, as well as an emotional stress for parents. The Ponseti method of clubfoot correction, consisting of serial manipulations and casting, is now the gold standard of treatment. It has traditionally been described using plaster of Paris (POP) above-knee casts; however, recently semi-rigid fiberglass softcast (SRF, 3M Scotchcast) has grown in popularity. There are currently no randomized controlled trials to prove its efficacy with respect to POP.

ELIGIBILITY:
Inclusion Criteria:

* congenital idiopathic clubfoot

Exclusion Criteria:

* positional equinovarus
* teratologic etiologies of clubfoot
* treatment started at another center
* refuse randomization
* do not understand English

Ages: 1 Week to 12 Weeks | Sex: All
Age Groups: Child
Enrollment: 30 (Actual)

PRIMARY OUTCOMES:
number of casts required to correct the clubfoot deformities | time required for the foot to be ready for a percutaneous tendo-achilles tenotomy (if necessary), or when dorsiflexion of the ankle greater than or equal to 15 degrees (Pirani=0) was achieved

SECONDARY OUTCOMES:
need for percutaneous tendo-achilles tenotomy
total time in casts (weeks)
ease of cast removal
time of cast removal | number of minutes required for each cast removal
method(s) of cast removal
other concerns about the casting material (e.g. appearance, weight, cleaning, water resistance), and complications relating to the casting material.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Howard, MD, Principal Investigator — IWK Health Centre
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Background] Dobbs MB, Morcuende JA, Gurnett CA, Ponseti IV. Treatment of idiopathic clubfoot: an historical review. Iowa Orthop J. 2000;20:59-64. PMID 10934626
- [Background] Altman DG, Schulz KF, Moher D, Egger M, Davidoff F, Elbourne D, Gotzsche PC, Lang T; CONSORT GROUP (Consolidated Standards of Reporting Trials). The revised CONSORT statement for reporting randomized trials: explanation and elaboration. Ann Intern Med. 2001 Apr 17;134(8):663-94. doi: 10.7326/0003-4819-134-8-200104170-00012. PMID 11304107
- [Background] Berman AT, Parks BG. A comparison of the mechanical properties of fiberglass cast materials and their clinical relevance. J Orthop Trauma. 1990;4(1):85-92. doi: 10.1097/00005131-199003000-00015. PMID 2313436
- [Background] Carroll NC. Clubfoot: what have we learned in the last quarter century? J Pediatr Orthop. 1997 Jan-Feb;17(1):1-2. No abstract available. PMID 8989690
- [Background] Colburn M, Williams M. Evaluation of the treatment of idiopathic clubfoot by using the Ponseti method. J Foot Ankle Surg. 2003 Sep-Oct;42(5):259-67. doi: 10.1016/s1067-2516(03)00312-0. PMID 14566717
- [Background] Cooper DM, Dietz FR. Treatment of idiopathic clubfoot. A thirty-year follow-up note. J Bone Joint Surg Am. 1995 Oct;77(10):1477-89. doi: 10.2106/00004623-199510000-00002. PMID 7593056
- [Background] Coss HS, Hennrikus WL. Parent satisfaction comparing two bandage materials used during serial casting in infants. Foot Ankle Int. 1996 Aug;17(8):483-6. doi: 10.1177/107110079601700809. PMID 8863028
- [Background] Dobbs MB, Corley CL, Morcuende JA, Ponseti IV. Late recurrence of clubfoot deformity: a 45-year followup. Clin Orthop Relat Res. 2003 Jun;(411):188-92. doi: 10.1097/01.blo.0000065837.77325.19. PMID 12782875
- [Background] Dobbs MB, Rudzki JR, Purcell DB, Walton T, Porter KR, Gurnett CA. Factors predictive of outcome after use of the Ponseti method for the treatment of idiopathic clubfeet. J Bone Joint Surg Am. 2004 Jan;86(1):22-7. doi: 10.2106/00004623-200401000-00005. PMID 14711941
- [Background] Flynn JM, Donohoe M, Mackenzie WG. An independent assessment of two clubfoot-classification systems. J Pediatr Orthop. 1998 May-Jun;18(3):323-7. PMID 9600557
- [Background] Haft GF, Walker CG, Crawford HA. Early clubfoot recurrence after use of the Ponseti method in a New Zealand population. J Bone Joint Surg Am. 2007 Mar;89(3):487-93. doi: 10.2106/JBJS.F.00169. PMID 17332096
- [Background] Herzenberg JE, Radler C, Bor N. Ponseti versus traditional methods of casting for idiopathic clubfoot. J Pediatr Orthop. 2002 Jul-Aug;22(4):517-21. PMID 12131451
- [Background] Ippolito E, Farsetti P, Caterini R, Tudisco C. Long-term comparative results in patients with congenital clubfoot treated with two different protocols. J Bone Joint Surg Am. 2003 Jul;85(7):1286-94. doi: 10.2106/00004623-200307000-00015. PMID 12851354
- [Background] Ippolito E, Fraracci L, Farsetti P, Di Mario M, Caterini R. The influence of treatment on the pathology of club foot. CT study at maturity. J Bone Joint Surg Br. 2004 May;86(4):574-80. PMID 15174556
- [Background] Laaveg SJ, Ponseti IV. Long-term results of treatment of congenital club foot. J Bone Joint Surg Am. 1980 Jan;62(1):23-31. PMID 7351412
- [Background] Mihalko WM, Beaudoin AJ, Krause WR. Mechanical properties and material characteristics of orthopaedic casting material. J Orthop Trauma. 1989;3(1):57-63. doi: 10.1097/00005131-198903010-00011. PMID 2709205
- [Background] Morcuende JA, Abbasi D, Dolan LA, Ponseti IV. Results of an accelerated Ponseti protocol for clubfoot. J Pediatr Orthop. 2005 Sep-Oct;25(5):623-6. doi: 10.1097/01.bpo.0000162015.44865.5e. PMID 16199943
- [Background] Noonan KJ, Richards BS. Nonsurgical management of idiopathic clubfoot. J Am Acad Orthop Surg. 2003 Nov-Dec;11(6):392-402. doi: 10.5435/00124635-200311000-00003. PMID 14686824
- [Background] Pirani S, Zeznik L, Hodges D. Magnetic resonance imaging study of the congenital clubfoot treated with the Ponseti method. J Pediatr Orthop. 2001 Nov-Dec;21(6):719-26. PMID 11675543
- [Background] Pittner DE, Klingele KE, Beebe AC. Treatment of clubfoot with the Ponseti method: a comparison of casting materials. J Pediatr Orthop. 2008 Mar;28(2):250-3. doi: 10.1097/BPO.0b013e318164f8e7. PMID 18388724
- [Background] Ponseti IV. The ponseti technique for correction of congenital clubfoot. J Bone Joint Surg Am. 2002 Oct;84(10):1889-90; author reply 1890-1. doi: 10.2106/00004623-200210000-00026. No abstract available. PMID 12377924
- [Background] Ponseti IV. Relapsing clubfoot: causes, prevention, and treatment. Iowa Orthop J. 2002;22:55-6. No abstract available. PMID 12180612
- [Background] Ponseti IV. Clubfoot management. J Pediatr Orthop. 2000 Nov-Dec;20(6):699-700. doi: 10.1097/00004694-200011000-00001. No abstract available. PMID 11097239
- [Background] Ponseti IV. Common errors in the treatment of congenital clubfoot. Int Orthop. 1997;21(2):137-41. doi: 10.1007/s002640050137. PMID 9195271
- [Background] Ponseti IV, Campos J. Observations on pathogenesis and treatment of congenital clubfoot. Clin Orthop Relat Res. 1972 May;84:50-60. doi: 10.1097/00003086-197205000-00011. No abstract available. PMID 5032850
- [Background] Ponseti IV. Treatment of congenital club foot. J Bone Joint Surg Am. 1992 Mar;74(3):448-54. No abstract available. PMID 1548277
- [Background] Roye DP Jr, Roye BD. Idiopathic congenital talipes equinovarus. J Am Acad Orthop Surg. 2002 Jul-Aug;10(4):239-48. doi: 10.5435/00124635-200207000-00002. PMID 15089073
- [Background] Silfverskiold JP. Fiberglass versus plaster casts. How to choose between them. Postgrad Med. 1989 Oct;86(5):71-2, 74. doi: 10.1080/00325481.1989.11704430. PMID 2636865
- [Background] Tindall AJ, Steinlechner CW, Lavy CB, Mannion S, Mkandawire N. Results of manipulation of idiopathic clubfoot deformity in Malawi by orthopaedic clinical officers using the Ponseti method: a realistic alternative for the developing world? J Pediatr Orthop. 2005 Sep-Oct;25(5):627-9. doi: 10.1097/01.bpo.0000164876.97949.6b. PMID 16199944
- [Background] Morcuende JA, Dolan LA, Dietz FR, Ponseti IV. Radical reduction in the rate of extensive corrective surgery for clubfoot using the Ponseti method. Pediatrics. 2004 Feb;113(2):376-80. doi: 10.1542/peds.113.2.376. PMID 14754952
- [Background] Ponseti I, Morcuende J, Mosca V, Pirani S, Dietz F, Herzenberg J, Weinstein S, Penny N, Michiel Steenbeek. Clubfoot: Ponseti Management Second Edition. Global-HELP publication
- See also: Website provides links to the publication entitled: Clubfoot: Ponseti Management — http://www.global-help.org